CLINICAL TRIAL: NCT02528357
Title: A Phase I, Open-Label Study of GSK3174998 Administered Alone and in Combination With Anticancer Agents Including Pembrolizumab in Subjects With Selected Advanced Solid Tumors
Brief Title: GSK3174998 Alone and With Pembrolizumab in Participants With Advanced Solid Tumors (ENGAGE-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201212; 2015-000152-14 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Neoplasms
Keywords: GSK3174998; Non-small Cell Lung Cancer (NSCLC); OX40; Pembrolizumab; Monoclonal Antibody (mAb); Selected Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Part 1A: GSK3174998 Monotherapy- Dose escalation (Experimental): Participants will receive GSK3174998 intravenously (IV) (dose range 0.003 to 10.0 milligram per kilogram [mg/kg]) every 3 weeks (Q3W) for up to 2 years or 35 cycles, whichever comes first.
  Interventions: Drug: GSK3174998
- Part 2A: GSK3174998+ pembrolizumab - Dose escalation (Experimental): Participants will receive GSK3174998 IV (dose range 0.003 to 10.0 mg/kg) Q3W for up to 2 years or 35 cycles, whichever comes first + Pembrolizumab 200 mg IV Q3W for up to 2 years or 35 cycles, whichever comes first.
  Interventions: Drug: GSK3174998; Drug: Pembrolizumab
- Part 2B: GSK3174998+ pembrolizumab - Cohort expansion (Experimental): Participants will receive GSK3174998 IV (at one dose level shown to be tolerable in dose escalation of part 2A) Q3W for up to 2 years or 35 cycles, whichever comes first + Pembrolizumab 200 mg IV Q3W for 2 years or 35 cycles, whichever comes first.
  Interventions: Drug: GSK3174998; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GSK3174998 — Lyophilized powder 40 mg reconstituted to get a dose range of 0.003 to <=10 mg/kg to be given as IV infusion for 30 minutes (min), Q3W
Drug: Pembrolizumab — Pembrolizumab as 100 mg/4 milliliter (mL) solution (dose: 200 mg) to be given as IV infusion for 30 min, Q3W
  Arms: Part 2A: GSK3174998+ pembrolizumab - Dose escalation; Part 2B: GSK3174998+ pembrolizumab - Cohort expansion

SUMMARY:
This is a first time in human (FTIH), open-label, non-randomized, multicenter study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary clinical activity of GSK3174998 administered intravenously to participants with selected advanced or recurrent solid tumors. This dose-escalation study will assess the safety, activity of GSK3174998 as monotherapy (Part 1), in combination with pembrolizumab (Part 2), and potentially in combination with additional therapies.

The study will be conducted in 2 parts, each part consisting of starting with a dose-escalation phase followed by a cohort expansion phase. GSK3174998 will first be evaluated as monotherapy in escalating doses. Once a dose of GSK3174998 has been identified that is both tolerable and demonstrates pharmacodynamic activity, enrollment of Part 2 may begin. In Part 2, escalating doses of GSK3174998 will be evaluated with fixed doses of pembrolizumab.

The maximum duration of treatment with GSK3174998 and pembrolizumab will be approximately 2 years or 35 cycles, whichever comes first. The follow-up period for safety assessments will be a minimum of 3 months from the date of the last dose. The post-treatment follow-up period will include disease assessments every 12 weeks until documented progressive disease (PD). Approximately 141 participants with selected advanced or recurrent solid tumors will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed, written informed consent.
* Male and female participants, age >=18 years (at the time consent is obtained).
* Histological documentation of locally advanced, recurrent or metastatic solid malignancy that has progressed after standard therapy appropriate for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate. Participants should not have received more than 5 prior lines of therapy for advanced disease including both standards of care and investigational therapies. Participants whose cancers harbor molecular alterations for which targeted therapy is standard of care should have received health authority approved appropriate targeted therapy for their tumor types before enrollment.
* Participants with the following solid tumors are eligible for screening: Non-small cell lung cancer (NSCLC), Squamous cell carcinoma of the head and neck (SCCHN), Renal cell carcinoma (RCC), melanoma, bladder, Soft Tissue Sarcoma (STS), Triple-negative breast cancer (TNBC), and Colorectal carcinoma displaying high microsatellite instability (MSI CRC). In Part 2B (Cohort Expansion), specific subgroups of the above solid tumors will be studied. These subgroups may be defined by specific lines of treatment, types of prior treatment, histological subtypes, and may be enriched for selected biomarkers or participant characteristics. Populations to be studied in Amendment 3 include but are not limited to the following. Enrolment of additional populations will be communicated in writing: Participants with dedifferentiated liposarcoma who have not received prior treatment with a Programmed death ligand 1 (PD-L1) inhibitor; Participants with melanoma who have received a prior PD-L1 inhibitor, had a CR, PR or SD and subsequently progressed while on PD-L1 therapy. Participants who have received prior treatment with a PD-L1 inhibitor must have documented disease progression as defined by meeting all of the following criteria: Has received at least 2 doses of an approved PD-L1 inhibitor; has demonstrated disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The initial evidence of disease progression is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD , in the absence of rapid clinical progression; Progressive disease has been documented within 18 weeks from the last dose of the PD-L1 inhibitor.
* In Parts 1A and 2A, a biopsy of the tumor tissue obtained at anytime from the initial diagnosis to study entry. Although a fresh biopsy obtained during screening is preferred, archival tumor specimen is acceptable if it is not feasible to obtain a fresh biopsy.

Participants enrolled in Part 1A or Part 2A Pharmacodynamic Cohorts or in Part 2B of the study must provide a fresh biopsy of a tumor lesion not previously irradiated during the screening period and must agree to provide at least one additional on-treatment biopsy. In addition, an archived tumor tissue should be submitted for Participants in Part 2B, if available. The criterion for collection of fresh biopsies may be waived once GlaxoSmithKline (GSK)has determined an appropriate number of viable tissue samples have been analyzed For Part 1B and Part 2B, any archival tumor specimen must have been obtained within 3 months of starting study drug.

* Measurable disease as per RECIST v1.1
* Palpable lesions that are not measurable by radiologic or photographic evaluations may not be utilized as the only measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Life expectancy of at least 12 weeks.
* Adequate organ function as defined by System Laboratory Values; Hematologic (Absolute neutrophil count [ANC] >=1.5x10^9/ liter [L], Lymphocyte count >=800/cubic millimeter [mm^3], Hemoglobin >=9 grams/deciliter [g/dL], Platelets >=100x10^9/L), Hepatic (Total bilirubin <=1.5x upper limit of normal [ULN] [For participants with Gilbert's Syndrome, only if direct bilirubin <=35 percent (%), <=3.0xULN], for Part 1A and 2A: alanine aminotransferase [ALT] <=1.5xULN), Part 2B: ALT <=2.5xULN; Renal (Serum Creatinine <=1.5xULN OR Calculated creatinine clearance [CrCl >50 mL/min ) and Endocrine (Thyroid stimulating hormone [TSH]) within normal limits. If TSH is not within normal limits at baseline, the participant may still be eligible if total triiodothyronine (T3) or free T3 and free thyroxine (T4) are within the normal limits.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec) or <480 msec for participants with bundle branch block.
* In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Female participant: is eligible to participate if she is not pregnant (as confirmed by a negative serum beta-human chorionic gonadotrophin [beta-hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion ; Hysterectomy; Documented Bilateral Oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

* Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until 120 days after the last dose of study medication and completion of the follow-up visit. GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP).

This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for participants who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis: Contraceptive subdermal implant with a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system with a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.

* Male Participants with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 120 days after the last dose of study medication: Vasectomy with documentation of azoospermia; Male condom plus partner use of one of the contraceptive options below; Contraceptive subdermal implant with a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system with a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.

Exclusion Criteria:

* Prior treatment with the following agents (from last dose of prior treatment to first dose of GSK3174998): Tumor necrosis factor receptor (TNFR) agonists, including OX40, CD27, CD137 (4-1BB), CD357 (GITR): at any time; Checkpoint inhibitors, including Programmed death receptor-1 (PD-1),

  1, and cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors: within 4 weeks; other anticancer therapy, including chemotherapy, targeted therapy, and biological therapy: within 4 weeks or 5 half lives of the drug, whichever is shorter. Prior radiation therapy is permissible if at least one unirradiated measurable lesion is available for assessment via RECIST version 1.1. A wash out of at least two weeks before start of study drug for palliative radiation to the extremities for osseous bone metastases and 4 weeks for radiation to the chest, brain, or visceral organs is required; Investigational therapy: if the participant has participated in a clinical trial and has received an investigational product: within 30 days or 5 half-lives of the investigational product (whichever is shorter). At least 14 days must have passed between the last dose of prior investigational agent and the first dose of study drug.
* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Toxicity from previous treatment: Participants with >=Grade 3 toxicity related to prior immunotherapy leading to study treatment discontinuation are not eligible; participants whose toxicity related to prior treatment has not resolved to <=Grade 1 (except alopecia, hearing loss, grade <=2 neuropathy or endocrinopathy managed with replacement therapy) are not eligible.
* Malignancy other than disease under study, except as noted below: any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the principal investigators and GSK Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on currently targeted malignancy, can be included in this clinical trial.
* Central nervous system (CNS) metastases, with the following exception: Participants who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids for 2 weeks prior to first dose of study drug.
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GMCSF], recombinant erythropoietin) within 2 weeks before the first dose of study drug.
* Major surgery <=4 weeks before the first dose of study treatment. Participants must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
* Active autoimmune disease that has required systemic treatment within the last 2 years (that is with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (example [e.g.], thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Concurrent medical condition requiring the use of systemic immunosuppressive medications within 28 days before the first dose of study treatment. Physiologic doses of corticosteroids for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids may be continued if the participant is on a stable dose.
* Active infection, known human immunodeficiency virus infection, or positive test for hepatitis B surface antigen or hepatitis C.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
* Known, current drug or alcohol abuse.
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
* Receipt of any live vaccine within 4 weeks.
* Recent history of allergen desensitization therapy within 4 weeks of starting study Treatment.
* History of severe hypersensitivity to other mAbs.
* History or evidence of cardiovascular risk including any of the following: Recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities including second degree (Type II) or third degree atrioventricular block; Documented cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrollment; documented congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system; recent (within the past 6 months) history of symptomatic pericarditis Current or history of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other condition that could interfere with the participant's safety, obtaining informed consent, or compliance to the study procedures.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific participant.
* History of severe hypersensitivity (>=Grade 3) to pembrolizumab and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Villejuif, France
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Postel-Vinay S, Lam VK, Ros W, Bauer TM, Hansen AR, Cho DC, Stephen Hodi F, Schellens JHM, Litton JK, Aspeslagh S, Autio KA, Opdam FL, McKean M, Somaiah N, Champiat S, Altan M, Spreafico A, Rahma O, Paul EM, Ahlers CM, Zhou H, Struemper H, Gorman SA, Watmuff M, Yablonski KM, Yanamandra N, Chisamore MJ, Schmidt EV, Hoos A, Marabelle A, Weber JS, Heymach JV. First-in-human phase I study of the OX40 agonist GSK3174998 with or without pembrolizumab in patients with selected advanced solid tumors (ENGAGE-1). J Immunother Cancer. 2023 Mar;11(3):e005301. doi: 10.1136/jitc-2022-005301. PMID 36927527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2 part study conducted across 4 countries. Part 1 was dose-escalation study to evaluate GSK3174998 monotherapy. Part 2 included dose-escalation cohorts of GSK3174998+pembrolizumab combination therapy (Comb. Th.) (Part 2A) and dose-expansion (Expan.) disease specific cohorts (Coh.) of GSK3174998 + pembrolizumab (Part 2B).
Pre-assignment Details: A total of 141 participants were enrolled in the study: 45 participants in Part 1 and 96 participants in Part 2 (74 in Part 2A+ 22 in Part 2B).
Groups:
- Part 1: GSK3174998 0.003 mg/kg: Participants received intravenous (IV) dose of GSK3174998 0.003 milligram per kilogram (mg/kg) every 3 weeks (wks) in Part 1.
- Part 1: GSK3174998 0.01 mg/kg: Participants received IV dose of GSK3174998 0.01 mg/kg every 3 weeks (Q3W) in Part 1.
- Part 1: GSK3174998 0.03 mg/kg: Participants received IV dose of GSK3174998 0.03 mg/kg Q3W in Part 1.
- Part 1: GSK3174998 0.1 mg/kg: Participants received IV dose of GSK3174998 0.1 mg/kg Q3W in Part 1.
- Part 1: GSK3174998 0.3 mg/kg: Participants received IV dose of GSK3174998 0.3 mg/kg Q3W in Part 1.
- Part 1: GSK3174998 1.0 mg/kg: Participants received IV dose of GSK3174998 1.0 mg/kg Q3W in Part 1.
- Part 1: GSK3174998 3.0 mg/kg: Participants received IV dose of GSK3174998 3.0 mg/kg Q3W in Part 1.
- Part 1: GSK3174998 10.0 mg/kg: Participants received IV dose of GSK3174998 10.0 mg/kg Q3W in Part 1.
- Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 0.003 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 0.01 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 0.03 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 0.1 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 0.3 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 1.0 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 3.0 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg: Participants received IV dose of GSK3174998 10.0 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2A.
- Part 2B: Melanoma Cohort: Participants with melanoma were included in this cohort and received IV dose of GSK3174998 0.3 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2B.
- Part 2B: Soft Tissue Sarcoma Cohort: Participants with soft tissue sarcoma were included in this cohort and received IV dose of GSK3174998 0.3 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2B.
- Part 2B: NSCLC Cohort: Participants with non-small cell lung cancer (NSCLC) were included in this cohort and received IV dose of GSK3174998 0.3 mg/kg + pembrolizumab 200 mg IV Q3W in Part 2B.
Period: Part1:Monotherapy(Up to Maximum 39weeks)
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Started | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 6 | 9 | 6 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 2 | 1 | 4 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Follow-up assessments removed (Protocol Amendment 4) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part2A:Comb. Th. (Up to Maximum 105wks)
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 7 | 9 | 9 | 6 | 5 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 5 | 6 | 7 | 0 | 0 | 0 | 0
Not completed — Investigator site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Follow-up assessments removed (Protocol Amendment 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Period: Part2B:Expan. Coh.(Up to Maximum 33 Wks)
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Follow-up assessments removed (Protocol Amendment 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort | Total
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4 | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4 | 9 | 8 | 5 | 141
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 1 | 0 | 5 | 8 | 4 | 2 | 4 | 2 | 1 | 3 | 6 | 6 | 8 | 6 | 6 | 1 | 6 | 5 | 2 | 76
  65 to 84 years | 0 | 1 | 3 | 2 | 6 | 2 | 3 | 2 | 4 | 2 | 4 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 3 | 64
  >=85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 6 | 6 | 5 | 1 | 6 | 3 | 3 | 3 | 8 | 5 | 6 | 3 | 8 | 0 | 3 | 4 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 2 | 4 | 5 | 3 | 1 | 1 | 2 | 2 | 2 | 7 | 8 | 9 | 4 | 4 | 6 | 4 | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American/African Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Asian - Central/South Asian Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Asian - East Asian Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Asian - South East Asian Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: White - Arabic/North African Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: White - White/Caucasian/European Heritage | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 6 | 7 | 10 | 4 | 7 | 3 | 5 | 5 | 10 | 12 | 12 | 7 | 10 | 2 | 9 | 6 | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Race: Missing | NA — Data not reported due to participant's confidentiality and privacy concerns | NA — Data not reported due to participant's confidentiality and privacy concerns | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Serious Adverse Event (SAE) and Non-serious Adverse Event (Non-SAE)
Description: An adverse event is any untoward medical occurrence in a participant or clinical investigation participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward medical occurrence that, at any dose: resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population consisted of all participants who received at least one dose of GSK3174998.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  Any SAE | 1 | 0 | 3 | 7 | 2 | 1 | 2 | 1
  Any non-SAE | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4

2. Primary Outcome: Part 2A: Number of Participants With Any SAE and Non-SAE
Description: as for outcome 1
Time Frame: Up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  Any SAE | 1 | 1 | 6 | 4 | 4 | 4 | 2 | 2
  Any non-SAE | 5 | 5 | 10 | 12 | 13 | 12 | 12 | 4

3. Primary Outcome: Part 2B: Number of Participants With Any SAE and Non-SAE
Description: as for outcome 1
Time Frame: Up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  Any SAE | 1 | 2 | 1
  Any non-SAE | 9 | 8 | 4

4. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: An adverse event was considered as DLT if it was considered by the investigator to be clinically relevant and attributed (definitely, probably or possibly) to study treatment, occurred within the first 28 days of the treatment, and met 1 of the following criteria: Hematologic: Febrile neutropenia, Grade4 neutropenia of >7days requiring Granulocyte colony-stimulating factor (G-CSF), Grade4 anemia of any duration, Grade4 thrombocytopenia of any duration or Grade3 thrombocytopenia with bleeding as described in National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE version 4). Non-hematologic: Grade4 toxicity, Grade3 toxicity that cannot be controlled within 3days, Ocular toxicity of >=Grade3 or of Grade2 requiring systemic steroids. Any other event results in permanent discontinuation of treatment during the first 4 weeks of treatment or any other event which in the judgment of the investigator and GlaxoSmithKline medical monitor is considered to be a DLT.
Time Frame: 28 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2A: Number of Participants With DLTs
Description: as for outcome 4
Time Frame: 28 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Part 2B: Number of Participants With DLTs
Description: as for outcome 4
Time Frame: 28 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Any Adverse Event Leading to Withdrawal (AELD) From the Study
Description: An adverse event is any untoward medical occurrence in a participant or clinical investigation participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with any adverse event leading to withdrawal from the study is presented.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 2A: Number of Participants With Any Adverse Event Leading to Withdrawal From the Study
Description: as for outcome 7
Time Frame: Up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

9. Primary Outcome: Part 2B: Number of Participants With Any Adverse Event Leading to Withdrawal From the Study
Description: as for outcome 7
Time Frame: Up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants | 0 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants With Dose Reductions or Delay
Description: Number of participants who had any dose reduction or dose delay (GSK3174998) due to any reason have been presented.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  Dose reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose delay | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

11. Primary Outcome: Part 2A: Number of Participants With Dose Reductions or Delay
Description: Number of participants who had any dose reduction or dose delay (GSK3174998) due to any reason have been presented.
Time Frame: Up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  Dose reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose delay | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 2B: Number of Participants With Dose Reductions or Delay
Description: Number of participants who had any dose reduction or dose delay (GSK3174998) due to any reason have been presented.
Time Frame: Up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  Dose reduction | 0 | 0 | 0
  Dose delay | 0 | 0 | 0

13. Primary Outcome: Part 1: Number of Participants With Any Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin (Hb), leukocyte count (leuko.), lymphocyte count (Lymph.), neutrophil count (Neutro.) and platelet count (PC). The laboratory parameters were graded according to NCI-CTCAE version 4. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  Hb decreased (anemia) | 1 | 0 | 7 | 6 | 5 | 3 | 0 | 1
  Hb increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Leuko. increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leuko. decreased | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Lymph. decreased | 0 | 0 | 5 | 3 | 6 | 1 | 5 | 3
  Lymph. increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutro. decreased | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  PC decreased | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0

14. Primary Outcome: Part 2A: Number of Participants With Any Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: Hb, leuko., Lymph., Neutro. and PC. The laboratory parameters were graded according to NCI-CTCAE version 4. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  Hb decreased (anemia) | 2 | 2 | 2 | 5 | 4 | 3 | 5 | 1
  Hb increased | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Leuko. increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leuko. decreased | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1
  Lymph. decreased | 2 | 2 | 5 | 2 | 6 | 4 | 3 | 2
  Lymph. increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neutro. decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  PC decreased | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0

15. Primary Outcome: Part 2B: Number of Participants With Any Grade Change From Baseline in Hematology Parameters
Description: as for outcome 14
Time Frame: Baseline (Day 1) and up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  Hb decreased (anemia) | 2 | 2 | 1
  Hb increased | 0 | 0 | 0
  Leuko. increased | 0 | 0 | 0
  Leuko. decreased | 1 | 0 | 0
  Lymph. decreased | 3 | 3 | 2
  Lymph. increased | 0 | 0 | 0
  Neutro. decreased | 0 | 0 | 0
  PC decreased | 1 | 1 | 1

16. Primary Outcome: Part 1: Number of Participants With Any Grade Change From Baseline in Liver Function Laboratory Parameters
Description: Blood samples were collected for the analysis of following liver function laboratory parameters: alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST) and bilirubin. The laboratory parameters were graded according to NCI-CTCAE version 4. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  ALT increased | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1
  ALP increased | 1 | 0 | 3 | 3 | 5 | 1 | 0 | 2
  AST increased | 0 | 0 | 3 | 5 | 1 | 2 | 3 | 3
  Bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

17. Primary Outcome: Part 2A: Number of Participants With Any Grade Change From Baseline in Liver Function Laboratory Parameters
Description: Blood samples were collected for the analysis of following liver function laboratory parameters: ALT, ALP, AST and bilirubin. The laboratory parameters were graded according to NCI-CTCAE version 4. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  ALT increased | 0 | 1 | 1 | 3 | 4 | 2 | 2 | 1
  ALP increased | 1 | 3 | 4 | 1 | 3 | 2 | 4 | 1
  AST increased | 1 | 3 | 2 | 1 | 6 | 3 | 3 | 1
  Bilirubin increased | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0

18. Primary Outcome: Part 2B: Number of Participants With Any Grade Change From Baseline in Liver Function Laboratory Parameters
Description: as for outcome 17
Time Frame: Baseline (Day 1) and up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  ALT increased | 2 | 0 | 0
  ALP increased | 3 | 4 | 0
  AST increased | 3 | 0 | 0
  Bilirubin increased | 1 | 0 | 0

19. Primary Outcome: Part 1: Number of Participants With Any Grade Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were graded using NCI-CTCAE version 4. For SBP: Grade 0: <120 millimeter mercury (mmHg); Grade 1: 120-139 mmHg; Grade 2: 140-159 mmHg; Grade 3: >=160 mmHg. For DBP: Grade 0: <80 mmHg; Grade 1: 80-89 mmHg; Grade 2: 90-99 mmHg; Grade 3: >=100 mmHg. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  SBP | 0 | 1 | 6 | 3 | 5 | 2 | 6 | 3
  DBP | 0 | 0 | 4 | 5 | 5 | 2 | 2 | 2

20. Primary Outcome: Part 2A: Number of Participants With Any Grade Change From Baseline in SBP and DBP
Description: SBP and DBP were graded using NCI-CTCAE version 4. For SBP: Grade 0: <120 mmHg; Grade 1: 120-139 mmHg; Grade 2: 140-159 mmHg; Grade 3: >=160 mmHg. For DBP: Grade 0: <80 mmHg; Grade 1: 80-89 mmHg; Grade 2: 90-99 mmHg; Grade 3: >=100 mmHg. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date (Day 1). Any grade increase is defined as an increase in NCI-CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented. Only those participants with any grade increase have been presented.
Time Frame: Baseline (Day 1) and up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  SBP | 2 | 4 | 8 | 6 | 6 | 7 | 7 | 1
  DBP | 1 | 4 | 7 | 6 | 6 | 5 | 4 | 0

21. Primary Outcome: Part 2B: Number of Participants With Any Grade Change From Baseline in SBP and DBP
Description: as for outcome 20
Time Frame: Baseline (Day 1) and up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  SBP | 7 | 4 | 4
  DBP | 5 | 5 | 3

22. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Heart Rate (HR)
Description: Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date (Day 1). Change from Baseline was defined as post Baseline value minus Baseline value. Number of participants with worst case change from Baseline in heart rate is presented. Data was categorized as: heart rate 'decrease to low', 'increase to high' and 'change to normal or no change'; where low HR: <60 beats per minute [bpm]', normal HR: 60 to 100 bpm and high HR: >100 bpm. If values were unchanged (example: increase to >100 bpm to increase to >100 bpm), or whose value became normal, were recorded in the 'change to normal or no change' category. Participants were counted twice if the participant had both 'decreased to low' and 'increased to high' during post Baseline, so the percentages might not add to 100%.
Time Frame: Baseline (Day 1) and up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  Decrease to low | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Change to normal or no change | 0 | 0 | 4 | 3 | 4 | 2 | 4 | 2
  Increase to high | 1 | 1 | 3 | 6 | 6 | 1 | 3 | 2

23. Primary Outcome: Part 2A: Number of Participants With Worst Case Change From Baseline in HR
Description: Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date (Day 1). Change from Baseline was defined as post Baseline value minus Baseline value. Number of participants with worst case change from Baseline in heart rate is presented. Data was categorized as: heart rate 'decrease to low', 'increase to high' and 'change to normal or no change'; where low HR: <60 bpm', normal HR: 60 to 100 bpm and high HR: >100 bpm. If values were unchanged (example: increase to >100 bpm to increase to >100 bpm), or whose value became normal, were recorded in the 'change to normal or no change' category. Participants were counted twice if the participant had both 'decreased to low' and 'increased to high' during post Baseline, so the percentages might not add to 100%.
Time Frame: Baseline (Day 1) and up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  Decrease to low | 0 | 0 | 1 | 3 | 4 | 1 | 3 | 0
  Change to normal or no change | 5 | 4 | 7 | 6 | 8 | 8 | 6 | 4
  Increase to high | 0 | 1 | 2 | 3 | 2 | 3 | 3 | 0

24. Primary Outcome: Part 2B: Number of Participants With Worst Case Change From Baseline in HR
Description: as for outcome 23
Time Frame: Baseline (Day 1) and up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  Decrease to low | 2 | 1 | 0
  Change to normal or no change | 4 | 3 | 5
  Increase to high | 3 | 4 | 0

25. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Body Temperature
Description: Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date (Day 1). Change from Baseline was defined as post Baseline value minus Baseline value. Number of participants with worst case change from Baseline in body temperature is presented. Data was categorized as: 'decrease to low', 'increase to high' and 'change to normal or no change'; where low body temperature: <=35 degrees Celsius, normal body temperature: 35 to 38 degrees Celsius and high body temperature: >=38 degrees Celsius. If values were unchanged (example: increase to >=38 degrees Celsius to increase to >=38 degrees Celsius), or whose value became normal, were recorded in the 'change to normal or no change' category. Participants were counted twice if the participant had both 'decreased to low' and 'increased to high' during post Baseline, so the percentages might not add to 100%.
Time Frame: Baseline (Day 1) and up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants
  Decrease to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change to normal or no change | 1 | 1 | 8 | 8 | 9 | 3 | 7 | 4
  Increase to high | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0

26. Primary Outcome: Part 2A: Number of Participants With Worst Case Change From Baseline in Body Temperature
Description: as for outcome 25
Time Frame: Baseline (Day 1) and up to maximum 105 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 10 | 12 | 14 | 12 | 12 | 4
Participants
  Decrease to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change to normal or no change | 4 | 5 | 10 | 11 | 12 | 12 | 12 | 4
  Increase to high | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0

27. Primary Outcome: Part 2B: Number of Participants With Worst Case Change From Baseline in Body Temperature
Description: as for outcome 25
Time Frame: Baseline (Day 1) and up to maximum 33 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Participants
  Decrease to low | 0 | 0 | 0
  Change to normal or no change | 9 | 8 | 5
  Increase to high | 0 | 0 | 0

28. Primary Outcome: Part 1: Number of Participants With Worst Case Post-Baseline Abnormal Clinically Significant Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was obtained after the participant had rested at least 10 minutes in a semi-recumbent or supine position during the study using ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with worst case post Baseline abnormal clinical significant ECG findings are presented.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Part 2A: Number of Participants With Worst Case Post-Baseline Abnormal Clinically Significant ECG Findings
Description: as for outcome 28
Time Frame: Up to maximum 105 weeks
Population: All Treated Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 4 | 3 | 10 | 10 | 12 | 10 | 11 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Part 2B: Number of Participants With Worst Case Post-Baseline Abnormal Clinically Significant ECG Findings
Description: as for outcome 28
Time Frame: Up to maximum 33 weeks
Population: All Treated Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 4 | 7 | 4
Participants | 0 | 0 | 0

31. Secondary Outcome: Part 1: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or a partial response (PR) as the Best Overall Response (BOR), as assessed by the investigator per Response Evaluation Criteria In Solid Tumors (RECIST) Version (v) 1.1 criteria. CR: Disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR: >=30 percent (%) decrease in tumor burden compared with Baseline in two observations at least 4 weeks apart.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Part 2A: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a confirmed CR or PR as the BOR, as assessed by the investigator per RECIST v 1.1 criteria. CR: Disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR: >=30% decrease in tumor burden compared with Baseline in two observations at least 4 weeks apart.
Time Frame: Up to maximum 105 weeks
Population: All Treated Population. The efficacy outputs were presented according to planned study treatment. One participant in Part 2A was planned for 0.01mg, but received 0.003mg at first dose in error. One participant in Part 2A was planned for 0.003mg, but received 0.3mg at first dose in error. Hence, 'N' for the 'Part 2A: GSK3174998 0.01 mg/kg+Pembrolizumab 200 mg' arm is greater than that for the Participant Flow.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 6 | 10 | 12 | 13 | 12 | 12 | 4
Percentage of participants | 0 | 17 | 0 | 25 | 8 | 8 | 0 | 0

33. Secondary Outcome: Part 2B: Objective Response Rate (ORR)
Description: as for outcome 32
Time Frame: Up to maximum 33 weeks
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Percentage of participants | 0 | 0 | 0

34. Secondary Outcome: Part 1: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR or PR at any time, plus stable disease (SD) >=12 weeks as assessed by the investigator per RECIST v 1.1 criteria. CR: Disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR: >=30% decrease in tumor burden compared with Baseline in two observations at least 4 weeks apart. SD: 30% decrease in tumor burden compared with Baseline cannot be established nor 20% increase compared with nadir.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Percentage of participants | 0 | 0 | 0 | 10 | 20 | 0 | 14 | 75

35. Secondary Outcome: Part 2A: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR or PR at any time, plus SD >=12 weeks as assessed by the investigator per RECIST v 1.1 criteria. CR: Disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR: >=30% decrease in tumor burden compared with Baseline in two observations at least 4 weeks apart. SD: 30% decrease in tumor burden compared with Baseline cannot be established nor 20% increase compared with nadir.
Time Frame: Up to maximum 105 weeks
Population: as for outcome 32
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 6 | 10 | 12 | 13 | 12 | 12 | 4
Percentage of participants | 0 | 33 | 0 | 50 | 23 | 50 | 58 | 0

36. Secondary Outcome: Part 2B: Disease Control Rate (DCR)
Description: as for outcome 35
Time Frame: Up to maximum 33 weeks
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Percentage of participants | 11 | 0 | 60

37. Secondary Outcome: Part 1: Plasma Concentrations of GSK3174998 at Indicated Time Points
Description: Blood samples for pharmacokinetic (PK) analysis of GSK3174998 were collected on Days 1, 22: Pre-dose and within 30 minutes, 4 hour, 24 hour after end of GSK3174998 infusion (EOI); anytime on Days 8, 15, 29 and 36; Days 43, 64, 85, 106: Pre-dose and within 30 minutes after end of GSK3174998 infusion.
Time Frame: Days 1, 22: Pre-dose and within 30 minutes, 4 hours, 24 hours after end of GSK3174998 infusion; anytime on Days 8,15,29,36; Days 43, 64, 85, 106: Pre-dose and within 30 minutes after end of GSK3174998 infusion
Population: Pharmacokinetic Population consisted of all participants from the All Treated Population for whom a PK sample was obtained and analyzed. Only those participants with data available at the indicated data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Micrograms per milliliter
  Day 1, predose, n=1,1,8,10,10,4,7,4 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (0.0000) | 0.001 (0.0033) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day1, 30minutes after EOI, n=1,1,8,10,10,4,7,4 | 0.044 (NA) — Standard deviation could not be calculated due to single participant | 0.181 (NA) — Standard deviation could not be calculated due to single participant | 0.893 (0.3505) | 2.958 (1.1359) | 6.091 (1.6075) | 23.224 (5.2813) | 77.500 (17.8619) | 277.615 (30.9564)
  Day1, 4hour after EOI, n=1,1,8,10,9,4,7,4: number analyzed (Participants) | 1 | 1 | 8 | 10 | 9 | 4 | 7 | 4
  Day1, 4hour after EOI, n=1,1,8,10,9,4,7,4 | 0.021 (NA) — Standard deviation could not be calculated due to single participant | 0.140 (NA) — Standard deviation could not be calculated due to single participant | 0.809 (0.3205) | 2.668 (1.0513) | 5.615 (1.3647) | 21.533 (5.5070) | 70.603 (15.1388) | 243.701 (42.5698)
  Day1, 24hour after EOI, n=1,1,6,10,9,4,7,4: number analyzed (Participants) | 1 | 1 | 6 | 10 | 9 | 4 | 7 | 4
  Day1, 24hour after EOI, n=1,1,6,10,9,4,7,4 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.083 (NA) — Standard deviation could not be calculated due to single participant | 0.564 (0.2508) | 2.080 (0.9446) | 4.954 (1.2600) | 17.645 (3.8210) | 59.143 (12.1864) | 191.862 (35.7293)
  Day 8, n=1,1,8,10,10,3,7,4: number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 3 | 7 | 4
  Day 8, n=1,1,8,10,10,3,7,4 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.122 (0.0926) | 0.678 (0.4251) | 1.932 (0.3732) | 9.675 (2.9619) | 32.974 (8.4840) | 108.278 (44.5563)
  Day 14, n=1,1,8,9,10,3,7,4: number analyzed (Participants) | 1 | 1 | 8 | 9 | 10 | 3 | 7 | 4
  Day 14, n=1,1,8,9,10,3,7,4 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.022 (0.0412) | 0.190 (0.1577) | 1.205 (0.2799) | 5.303 (1.9430) | 21.705 (6.4334) | 80.909 (27.3394)
  Day 22, predose, n=1,1,8,10,10,4,7,4 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.003 (0.0087) | 0.026 (0.0529) | 0.605 (0.2412) | 2.826 (2.1396) | 15.185 (4.1187) | 58.537 (17.2736)
  Day22, 30minutes after EOI, n=1,1,8,10,10,4,7,4 | 0.043 (NA) — Standard deviation could not be calculated due to single participant | 0.174 (NA) — Standard deviation could not be calculated due to single participant | 0.619 (0.2229) | 2.579 (0.4762) | 7.256 (1.8199) | 25.859 (9.2995) | 81.115 (32.5472) | 321.132 (40.4375)
  Day22, 4hour after EOI, n=1,1,8,10,9,4,7,4: number analyzed (Participants) | 1 | 1 | 8 | 10 | 9 | 4 | 7 | 4
  Day22, 4hour after EOI, n=1,1,8,10,9,4,7,4 | 0.038 (NA) — Standard deviation could not be calculated due to single participant | 0.149 (NA) — Standard deviation could not be calculated due to single participant | 0.523 (0.1963) | 2.301 (0.4088) | 6.519 (1.5717) | 22.905 (9.6502) | 82.690 (18.1793) | 306.585 (31.7702)
  Day22, 24hour after EOI, n=1,0,6,9,9,4,7,4: number analyzed (Participants) | 1 | 0 | 6 | 9 | 9 | 4 | 7 | 4
  Day22, 24hour after EOI, n=1,0,6,9,9,4,7,4 | 0.012 (NA) — Standard deviation could not be calculated due to single participant |  | 0.319 (0.1676) | 1.711 (0.4435) | 4.933 (0.8727) | 17.869 (9.3910) | 72.801 (17.5925) | 260.830 (44.1526)
  Day 29, n=0,1,8,10,10,4,7,4: number analyzed (Participants) | 0 | 1 | 8 | 10 | 10 | 4 | 7 | 4
  Day 29, n=0,1,8,10,10,4,7,4 |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.037 (0.0663) | 0.380 (0.2882) | 2.243 (0.8667) | 8.654 (5.9929) | 42.013 (13.3448) | 153.655 (37.5871)
  Day 36, n=0,1,7,9,9,4,6,4: number analyzed (Participants) | 0 | 1 | 7 | 9 | 9 | 4 | 6 | 4
  Day 36, n=0,1,7,9,9,4,6,4 |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.013 (0.0313) | 0.115 (0.1114) | 1.227 (0.4101) | 6.428 (4.5933) | 31.093 (10.5909) | 111.545 (22.8298)
  Day 43, predose, n=0,1,6,8,9,4,5,3: number analyzed (Participants) | 0 | 1 | 6 | 8 | 9 | 4 | 5 | 3
  Day 43, predose, n=0,1,6,8,9,4,5,3 |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.003 (0.0064) | 0.023 (0.0355) | 0.832 (0.5269) | 4.789 (3.2591) | 21.658 (8.9413) | 82.723 (26.1829)
  Day43, 30minutes after EOI, n=0,1,6,7,9,3,5,3: number analyzed (Participants) | 0 | 1 | 6 | 7 | 9 | 3 | 5 | 3
  Day43, 30minutes after EOI, n=0,1,6,7,9,3,5,3 |  | 0.267 (NA) — Standard deviation could not be calculated due to single participant | 0.547 (0.5929) | 2.130 (1.4403) | 7.373 (2.3810) | 30.602 (0.6521) | 95.775 (22.9300) | 302.882 (3.7341)
  Day 64, predose, n=0,1,5,5,7,4,4,3: number analyzed (Participants) | 0 | 1 | 5 | 5 | 7 | 4 | 4 | 3
  Day 64, predose, n=0,1,5,5,7,4,4,3 |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.023 (0.0520) | 0.014 (0.0206) | 1.097 (0.4744) | 5.747 (3.8915) | 23.922 (9.6447) | 76.602 (27.6046)
  Day64, 30minutes after EOI, n=0,0,5,5,7,4,4,2: number analyzed (Participants) | 0 | 0 | 5 | 5 | 7 | 4 | 4 | 2
  Day64, 30minutes after EOI, n=0,0,5,5,7,4,4,2 |  |  | 0.339 (0.4499) | 1.154 (1.2985) | 7.952 (2.7538) | 21.941 (15.0801) | 98.410 (19.0269) | 312.277 (61.0388)
  Day 85, predose, n=0,0,1,4,3,2,2,3: number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 2 | 2 | 3
  Day 85, predose, n=0,0,1,4,3,2,2,3 |  |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.023 (0.0315) | 1.227 (0.7462) | 8.518 (0.6700) | 22.635 (3.1816) | 83.090 (31.8311)
  Day85, 30minutes after EOI, n=0,0,1,4,3,2,2,3: number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 2 | 2 | 3
  Day85, 30minutes after EOI, n=0,0,1,4,3,2,2,3 |  |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 1.246 (1.3975) | 9.421 (1.8598) | 32.824 (0.4611) | 82.402 (18.5192) | 294.788 (15.9947)
  Day106, predose, n=0,0,1,1,2,2,1,2: number analyzed (Participants) | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2
  Day106, predose, n=0,0,1,1,2,2,1,2 |  |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 1.323 (0.2234) | 8.497 (0.5922) | 19.047 (NA) — Standard deviation could not be calculated due to single participant | 94.359 (11.4639)
  Day106, 30minutes after EOI, n=0,0,0,1,3,2,1,2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 2
  Day106, 30minutes after EOI, n=0,0,0,1,3,2,1,2 |  |  |  | 1.591 (NA) — Standard deviation could not be calculated due to single participant | 8.377 (0.3270) | 33.406 (6.3673) | 79.852 (NA) — Standard deviation could not be calculated due to single participant | 307.222 (3.5048)

38. Secondary Outcome: Part 2A: Plasma Concentrations of GSK3174998 at Indicated Time Points
Description: Blood samples for PK analysis of GSK3174998 were collected on Days 1, 22: Pre-dose and within 30 minutes, 4 hour, 24 hour after end of GSK3174998 infusion (EOI); anytime on Days 8, 15, 29 and 36; Days 43, 64, 85, 106: Pre-dose and within 30 minutes after end of GSK3174998 infusion.
Time Frame: as for outcome 37
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 4 | 5 | 10 | 11 | 14 | 11 | 12 | 4
Micrograms per milliliter
  Day 1, predose, n=4,5,9,10,11,11,12,4: number analyzed (Participants) | 4 | 5 | 9 | 10 | 11 | 11 | 12 | 4
  Day 1, predose, n=4,5,9,10,11,11,12,4 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.928 (3.0764) | 0.000 (0.0000) | 0.000 (0.0000)
  Day1, 30minutes after EOI, n=4,5,9,10,11,11,12,4: number analyzed (Participants) | 4 | 5 | 9 | 10 | 11 | 11 | 12 | 4
  Day1, 30minutes after EOI, n=4,5,9,10,11,11,12,4 | 0.051 (0.0212) | 0.235 (0.0971) | 0.833 (0.5313) | 2.088 (0.8049) | 6.542 (2.1648) | 25.623 (6.4576) | 70.550 (16.4984) | 193.082 (30.6483)
  Day1, 4hour after EOI, n=4,5,9,10,11,11,12,4: number analyzed (Participants) | 4 | 5 | 9 | 10 | 11 | 11 | 12 | 4
  Day1, 4hour after EOI, n=4,5,9,10,11,11,12,4 | 0.038 (0.0263) | 0.215 (0.0396) | 0.762 (0.4730) | 2.160 (1.0232) | 5.819 (1.6015) | 23.367 (4.5233) | 66.831 (17.5167) | 178.023 (20.6597)
  Day1, 24hour after EOI, n=4,5,9,10,11,11,12,4: number analyzed (Participants) | 4 | 5 | 9 | 10 | 11 | 11 | 12 | 4
  Day1, 24hour after EOI, n=4,5,9,10,11,11,12,4 | 0.010 (0.0125) | 0.112 (0.0599) | 0.578 (0.4049) | 1.644 (0.7086) | 5.084 (1.7161) | 19.398 (5.6732) | 55.782 (13.0007) | 140.747 (9.5100)
  Day 8, n=4,5,10,11,14,11,12,4 | 0.000 (0.0000) | 0.000 (0.0000) | 0.428 (0.9836) | 0.592 (0.3233) | 2.203 (0.7619) | 12.151 (8.5380) | 30.442 (8.6063) | 71.830 (14.1731)
  Day 15, n=4,4,10,10,12,11,12,4: number analyzed (Participants) | 4 | 4 | 10 | 10 | 12 | 11 | 12 | 4
  Day 15, n=4,4,10,10,12,11,12,4 | 0.000 (0.0000) | 0.000 (0.0000) | 0.257 (0.7547) | 0.200 (0.1821) | 1.357 (0.7574) | 8.458 (8.3133) | 22.050 (6.8631) | 50.342 (12.5709)
  Day 22, predose, n=3,2,10,10,12,10,12,3: number analyzed (Participants) | 3 | 2 | 10 | 10 | 12 | 10 | 12 | 3
  Day 22, predose, n=3,2,10,10,12,10,12,3 | 0.000 (0.0000) | 0.000 (0.0000) | 0.106 (0.3359) | 0.080 (0.0880) | 0.626 (0.3716) | 6.912 (7.0973) | 16.354 (5.5789) | 31.882 (12.4466)
  Day22, 30minutes after EOI, n=3,2,10,10,12,9,12,3: number analyzed (Participants) | 3 | 2 | 10 | 10 | 12 | 9 | 12 | 3
  Day22, 30minutes after EOI, n=3,2,10,10,12,9,12,3 | 0.080 (0.0350) | 0.879 (0.8898) | 0.754 (0.4533) | 2.343 (0.5196) | 7.496 (2.7519) | 30.238 (4.8782) | 85.882 (16.2709) | 222.118 (45.7084)
  Day22, 4hour after EOI, n=3,2,9,10,12,9,12,3: number analyzed (Participants) | 3 | 2 | 9 | 10 | 12 | 9 | 12 | 3
  Day22, 4hour after EOI, n=3,2,9,10,12,9,12,3 | 0.052 (0.0406) | 0.682 (0.6743) | 0.704 (0.4011) | 2.203 (0.4515) | 6.938 (2.6934) | 27.273 (6.0059) | 82.796 (16.8542) | 205.085 (26.1667)
  Day22, 24hour after EOI, n=3,2,7,7,9,10,12,3: number analyzed (Participants) | 3 | 2 | 7 | 7 | 9 | 10 | 12 | 3
  Day22, 24hour after EOI, n=3,2,7,7,9,10,12,3 | 0.011 (0.0188) | 0.365 (0.3729) | 0.628 (0.3755) | 1.702 (0.3438) | 6.015 (2.6501) | 21.631 (8.6914) | 69.978 (13.9446) | 164.798 (36.7704)
  Day 29, n=3,1,9,10,10,10,12,1: number analyzed (Participants) | 3 | 1 | 9 | 10 | 10 | 10 | 12 | 1
  Day 29, n=3,1,9,10,10,10,12,1 | 0.000 (0.0000) | 0.045 (NA) — Standard deviation could not be calculated due to single participant | 0.134 (0.2410) | 0.607 (0.3352) | 2.682 (1.5569) | 11.961 (5.5511) | 45.527 (14.7008) | 67.369 (NA) — Standard deviation could not be calculated due to single participant
  Day 36, n=3,2,8,8,8,10,11,1: number analyzed (Participants) | 3 | 2 | 8 | 8 | 8 | 10 | 11 | 1
  Day 36, n=3,2,8,8,8,10,11,1 | 0.000 (0.0000) | 0.000 (0.0000) | 0.019 (0.0404) | 0.243 (0.2081) | 1.994 (1.2562) | 9.146 (4.7873) | 33.671 (10.9055) | 106.605 (NA) — Standard deviation could not be calculated due to single participant
  Day 43, predose, n=3,3,7,7,8,9,12,1: number analyzed (Participants) | 3 | 3 | 7 | 7 | 8 | 9 | 12 | 1
  Day 43, predose, n=3,3,7,7,8,9,12,1 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.071 (0.1213) | 0.950 (0.6068) | 7.207 (2.1852) | 24.578 (8.5351) | 74.088 (NA) — Standard deviation could not be calculated due to single participant
  Day43, 30minutes after EOI, n=3,3,7,7,8,8,12,1: number analyzed (Participants) | 3 | 3 | 7 | 7 | 8 | 8 | 12 | 1
  Day43, 30minutes after EOI, n=3,3,7,7,8,8,12,1 | 0.071 (0.0156) | 0.229 (0.0379) | 0.496 (0.2657) | 1.922 (0.8919) | 7.639 (2.1641) | 28.433 (5.1446) | 94.463 (20.9570) | 377.078 (NA) — Standard deviation could not be calculated due to single participant
  Day 64, predose, n=1,3,2,6,4,8,10,0: number analyzed (Participants) | 1 | 3 | 2 | 6 | 4 | 8 | 10 | 0
  Day 64, predose, n=1,3,2,6,4,8,10,0 | 0.000 (NA) — Standard deviation could not be calculated due to single participant | 0.000 (0.0000) | 0.000 (0.0000) | 0.067 (0.1145) | 0.706 (0.8655) | 8.349 (2.7499) | 32.716 (11.1159) |
  Day64, 30minutes after EOI, n=1,3,2,7,4,8,10,0: number analyzed (Participants) | 1 | 3 | 2 | 7 | 4 | 8 | 10 | 0
  Day64, 30minutes after EOI, n=1,3,2,7,4,8,10,0 | 0.067 (NA) — Standard deviation could not be calculated due to single participant | 0.245 (0.0932) | 0.284 (0.4014) | 2.152 (1.3890) | 6.032 (3.2357) | 33.382 (5.0217) | 99.623 (25.2220) |
  Day 85, predose, n=0,3,0,5,5,7,8,0: number analyzed (Participants) | 0 | 3 | 0 | 5 | 5 | 7 | 8 | 0
  Day 85, predose, n=0,3,0,5,5,7,8,0 |  | 0.000 (0.0000) |  | 0.115 (0.1528) | 0.938 (0.9332) | 10.323 (3.5051) | 35.166 (13.8402) |
  Day85, 30minutes after EOI, n=0,3,0,5,5,7,8,0: number analyzed (Participants) | 0 | 3 | 0 | 5 | 5 | 7 | 8 | 0
  Day85, 30minutes after EOI, n=0,3,0,5,5,7,8,0 |  | 0.228 (0.0996) |  | 2.275 (1.2464) | 7.734 (2.5853) | 34.982 (6.5978) | 100.514 (26.7950) |
  Day106, predose, n=0,1,0,5,5,5,8,0: number analyzed (Participants) | 0 | 1 | 0 | 5 | 5 | 5 | 8 | 0
  Day106, predose, n=0,1,0,5,5,5,8,0 |  | 0.000 (NA) — Standard deviation could not be calculated due to single participant |  | 0.184 (0.1858) | 0.647 (0.8249) | 10.395 (5.5838) | 36.990 (16.0967) |
  Day106, 30minutes after EOI, n=0,1,0,5,4,5,8,0: number analyzed (Participants) | 0 | 1 | 0 | 5 | 4 | 5 | 8 | 0
  Day106, 30minutes after EOI, n=0,1,0,5,4,5,8,0 |  | 0.269 (NA) — Standard deviation could not be calculated due to single participant |  | 2.477 (0.8254) | 8.218 (3.9343) | 33.183 (6.7012) | 108.103 (29.3324) |

39. Secondary Outcome: Part 2B: Plasma Concentrations of GSK3174998 at Indicated Time Points
Description: as for outcome 38
Time Frame: as for outcome 37
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 4
Micrograms per milliliter
  Day 1, predose, n=7,5,3: number analyzed (Participants) | 7 | 5 | 3
  Day 1, predose, n=7,5,3 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day1, 30minutes after EOI, n=7,6,4: number analyzed (Participants) | 7 | 6 | 4
  Day1, 30minutes after EOI, n=7,6,4 | 6.132 (2.6768) | 5.668 (1.1752) | 7.618 (0.6794)
  Day1, 4hour after EOI, n=7,6,4: number analyzed (Participants) | 7 | 6 | 4
  Day1, 4hour after EOI, n=7,6,4 | 5.229 (2.1553) | 5.383 (0.6932) | 6.638 (1.2259)
  Day1, 24hour after EOI, n=7,5,0: number analyzed (Participants) | 7 | 5 | 0
  Day1, 24hour after EOI, n=7,5,0 | 4.000 (1.7095) | 4.141 (1.0168) |
  Day 8, n=8,7,4: number analyzed (Participants) | 8 | 7 | 4
  Day 8, n=8,7,4 | 1.972 (0.3899) | 2.062 (0.7993) | 2.501 (0.6042)
  Day 15, n=8,7,4: number analyzed (Participants) | 8 | 7 | 4
  Day 15, n=8,7,4 | 0.989 (0.3362) | 1.223 (0.5792) | 1.252 (0.3432)
  Day 22, predose, n=8,7,4: number analyzed (Participants) | 8 | 7 | 4
  Day 22, predose, n=8,7,4 | 0.401 (0.3015) | 0.646 (0.5756) | 0.444 (0.2856)
  Day22, 30minutes after EOI, n=8,7,4: number analyzed (Participants) | 8 | 7 | 4
  Day22, 30minutes after EOI, n=8,7,4 | 5.805 (0.8298) | 6.259 (1.3552) | 7.226 (0.8588)
  Day22, 4hour after EOI, n=8,7,4: number analyzed (Participants) | 8 | 7 | 4
  Day22, 4hour after EOI, n=8,7,4 | 5.722 (1.5376) | 5.810 (1.4074) | 7.363 (1.0038)
  Day22, 24hour after EOI, n=4,2,4: number analyzed (Participants) | 4 | 2 | 4
  Day22, 24hour after EOI, n=4,2,4 | 4.531 (0.6357) | 2.070 (0.5224) | 5.850 (1.3604)
  Day 29, n=9,8,4 | 1.715 (0.8979) | 2.201 (1.4063) | 2.070 (0.9160)
  Day 36, n=7,6,4: number analyzed (Participants) | 7 | 6 | 4
  Day 36, n=7,6,4 | 0.871 (0.7222) | 1.597 (1.2560) | 1.124 (0.5805)
  Day 43, predose, n=8,4,2: number analyzed (Participants) | 8 | 4 | 2
  Day 43, predose, n=8,4,2 | 0.442 (0.4862) | 1.045 (1.0289) | 0.570 (0.6971)
  Day43, 30minutes after EOI, n=8,4,2: number analyzed (Participants) | 8 | 4 | 2
  Day43, 30minutes after EOI, n=8,4,2 | 6.657 (1.1060) | 7.271 (2.0499) | 6.913 (2.3366)
  Day 64, predose, n=4,3,2: number analyzed (Participants) | 4 | 3 | 2
  Day 64, predose, n=4,3,2 | 0.726 (0.7935) | 1.520 (1.2083) | 0.663 (0.8153)
  Day64, 30minutes after EOI, n=4,3,2: number analyzed (Participants) | 4 | 3 | 2
  Day64, 30minutes after EOI, n=4,3,2 | 7.496 (1.7948) | 7.480 (2.0226) | 8.172 (0.5517)
  Day 85, predose, n=2,3,2: number analyzed (Participants) | 2 | 3 | 2
  Day 85, predose, n=2,3,2 | 0.976 (0.9973) | 1.631 (1.5426) | 0.711 (0.5122)
  Day85, 30minutes after EOI, n=2,3,2: number analyzed (Participants) | 2 | 3 | 2
  Day85, 30minutes after EOI, n=2,3,2 | 10.245 (0.2669) | 8.920 (2.4241) | 9.208 (1.3270)
  Day106, predose, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  Day106, predose, n=1,2,2 | 1.714 (NA) — Standard deviation could not be calculated due to single participant | 0.800 (1.0858) | 1.015 (0.6750)
  Day106, 30minutes after EOI, n=2,2,1: number analyzed (Participants) | 2 | 2 | 1
  Day106, 30minutes after EOI, n=2,2,1 | 9.933 (1.9969) | 6.324 (1.9856) | 8.673 (NA) — Standard deviation could not be calculated due to single participant

40. Secondary Outcome: Part 1: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) of GSK3174998
Description: Blood samples for PK analysis of GSK3174998 were collected on Days 1, 22: Pre-dose and within 30 minutes, 4 hour, 24 hour after end of GSK3174998 infusion; anytime on Days 8, 15, 29 and 36; Day 43: Pre-dose and within 30 minutes after end of GSK3174998 infusion. Each dosing cycle was of 21 days. PK parameters of GSK3174998 were calculated using non-compartmental methods.
Time Frame: Days 1, 22: Pre-dose and within 30 minutes, 4 hours, 24 hours after end of GSK3174998 infusion; anytime on Days 8,15,29,36; Day 43: Pre-dose and within 30 minutes after end of GSK3174998 infusion (each dosing cycle was of 21 days)
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed (represented by n=X in category titles). There were not enough samples with concentrations above lower limit of quantification to allow calculation of AUC(0-tau) for 0.003mg and 0.01mg arms in Cycles 1 and 2. There was not enough PK sampling in Cycles 3,4 and 5 for all arms to allow calculation of AUC(0-tau).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 6 | 10 | 9 | 3 | 7 | 4
Day*micrograms per milliliter
  Cycle 1, n=0,0,6,10,9,3,7,4 |  |  | 2.9362 (56.6) | 11.272 (57.8) | 39.374 (17.5) | 175.09 (33.2) | 630.94 (23.7) | 2129.9 (30.4)
  Cycle 2, n=0,0,2,7,9,2,4,3: number analyzed (Participants) | 0 | 0 | 2 | 7 | 9 | 2 | 4 | 3
  Cycle 2, n=0,0,2,7,9,2,4,3 |  |  | 2.2804 (102.7) | 8.7296 (62.8) | 46.093 (30.7) | 255.78 (12.5) | 866.23 (33.5) | 2859.4 (16.7)

41. Secondary Outcome: Part 2A: AUC(0-tau) of GSK3174998
Description: as for outcome 40
Time Frame: as for outcome 40
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed (represented by n=X in category titles). There were not enough samples with concentrations above lower limit of quantification to allow calculation of AUC(0-tau) for 0.003mg and 0.01mg arms in Cycles 1 and 2. There was not enough PK sampling in Cycles 3,4 and 5 in all arms to allow calculation of AUC(0-tau).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 4 | 10 | 9 | 8 | 12 | 3
Day*micrograms per milliliter
  Cycle 1, n=0,0,4,10,9,8,12,3 |  |  | 4.2333 (77.9) | 11.592 (42.4) | 40.936 (34.2) | 175.17 (32.6) | 605.22 (29.2) | 1465.8 (20.3)
  Cycle 2, n=0,0,2,6,7,8,12,1: number analyzed (Participants) | 0 | 0 | 2 | 6 | 7 | 8 | 12 | 1
  Cycle 2, n=0,0,2,6,7,8,12,1 |  |  | 4.0512 (64.9) | 10.862 (44.0) | 52.517 (78.9) | 271.67 (30.0) | 862.97 (30.8) | 2801.8 (NA) — Geometric coefficient of variation could not be calculated due to single participant

42. Secondary Outcome: Part 2B: AUC(0-tau) of GSK3174998
Description: as for outcome 40
Time Frame: as for outcome 40
Population: as for outcome 41
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 7 | 6 | 4
Day*micrograms per milliliter
  Cycle 1, n=7,6,4 | 38.781 (9.6) | 38.171 (43.4) | 46.544 (21.9)
  Cycle 2, n=7,4,2: number analyzed (Participants) | 7 | 4 | 2
  Cycle 2, n=7,4,2 | 39.504 (31.6) | 41.838 (96.8) | 33.502 (57.0)

43. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of GSK3174998
Description: Blood samples for PK analysis of GSK3174998 were collected on Days 1, 22: Pre-dose and within 30 minutes, 4 hour, 24 hour after end of GSK3174998 infusion; anytime on Days 8, 15, 29 and 36; Days 43, 64, 85, 106: Pre-dose and within 30 minutes after end of GSK3174998 infusion. Each dosing cycle was of 21 days. PK parameters of GSK3174998 were calculated using non-compartmental methods.
Time Frame: Days 1, 22: Pre-dose and within 30 minutes, 4 hours, 24 hours after end of GSK3174998 infusion; anytime on Days 8,15,29,36; Days 43, 64, 85, 106: Pre-dose and within 30 minutes after end of GSK3174998 infusion (each dosing cycle was of 21 days)
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Micrograms per milliliter
  Cmax, Cycle 1, n=1,1,8,10,10,4,7,4 | 0.04440 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.1814 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.8408 (43.1) | 2.808 (35.5) | 6.002 (24.0) | 22.70 (26.0) | 75.81 (22.9) | 276.4 (10.7)
  Cmax, Cycle 2, n=1,1,8,10,10,4,6,4: number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 6 | 4
  Cmax, Cycle 2, n=1,1,8,10,10,4,6,4 | 0.04280 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.1737 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.5816 (40.9) | 2.539 (20.4) | 7.096 (25.8) | 24.13 (49.4) | 90.26 (21.9) | 320.2 (12.1)
  Cmax, Cycle 3, n=0,1,6,7,9,3,5,3: number analyzed (Participants) | 0 | 1 | 6 | 7 | 9 | 3 | 5 | 3
  Cmax, Cycle 3, n=0,1,6,7,9,3,5,3 |  | 0.2671 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.2532 (369.2) | 1.355 (206.1) | 7.011 (35.7) | 30.60 (2.1) | 93.67 (23.7) | 302.9 (1.2)
  Cmax, Cycle 4, n=0,0,3,4,7,4,4,2: number analyzed (Participants) | 0 | 0 | 3 | 4 | 7 | 4 | 4 | 2
  Cmax, Cycle 4, n=0,0,3,4,7,4,4,2 |  |  | 0.3112 (395.0) | 0.5338 (1632.6) | 7.573 (34.5) | 8.117 (2535.5) | 97.02 (19.7) | 309.3 (19.9)
  Cmax, Cycle 5, n=0,0,0,3,3,2,2,3: number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 2 | 2 | 3
  Cmax, Cycle 5, n=0,0,0,3,3,2,2,3 |  |  |  | 1.024 (264.9) | 9.292 (20.9) | 32.82 (1.4) | 81.35 (23.0) | 294.5 (5.5)
  Cmin, Cycle 1, n=0,0,1,4,10,3,7,4: number analyzed (Participants) | 0 | 0 | 1 | 4 | 10 | 3 | 7 | 4
  Cmin, Cycle 1, n=0,0,1,4,10,3,7,4 |  |  | 0.02450 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.04138 (139.4) | 0.5417 (62.6) | 3.626 (35.4) | 14.73 (26.9) | 56.29 (34.8)
  Cmin, Cycle 2, n=0,0,1,3,9,3,5,3: number analyzed (Participants) | 0 | 0 | 1 | 3 | 9 | 3 | 5 | 3
  Cmin, Cycle 2, n=0,0,1,3,9,3,5,3 |  |  | 0.01570 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.05811 (50.0) | 0.6702 (86.3) | 6.353 (12.3) | 19.92 (51.3) | 79.63 (36.0)
  Cmin, Cycle 3, n=0,0,1,2,7,3,4,3: number analyzed (Participants) | 0 | 0 | 1 | 2 | 7 | 3 | 4 | 3
  Cmin, Cycle 3, n=0,0,1,2,7,3,4,3 |  |  | 0.1162 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.03436 (39.2) | 0.9979 (52.7) | 7.633 (10.9) | 22.57 (40.3) | 72.89 (41.5)
  Cmin, Cycle 4, n=0,0,0,2,3,2,2,3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 3
  Cmin, Cycle 4, n=0,0,0,2,3,2,2,3 |  |  |  | 0.04153 (75.0) | 1.053 (81.8) | 8.504 (7.9) | 22.52 (14.2) | 78.37 (45.9)
  Cmin, Cycle 5, n=0,0,0,0,2,2,1,2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2
  Cmin, Cycle 5, n=0,0,0,0,2,2,1,2 |  |  |  |  | 1.313 (17.1) | 8.486 (7.0) | 19.05 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 94.01 (12.2)

44. Secondary Outcome: Part 2A: Cmax and Cmin of GSK3174998
Description: as for outcome 43
Time Frame: as for outcome 43
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 4 | 5 | 9 | 10 | 12 | 9 | 12 | 4
Micrograms per milliliter
  Cmax, Cycle 1, n=4,5,9,10,11,9,12,4: number analyzed (Participants) | 4 | 5 | 9 | 10 | 11 | 9 | 12 | 4
  Cmax, Cycle 1, n=4,5,9,10,11,9,12,4 | 0.05321 (37.3) | 0.2505 (23.6) | 0.6748 (95.1) | 2.446 (23.4) | 6.345 (30.8) | 23.84 (18.9) | 71.37 (24.1) | 191.3 (16.0)
  Cmax, Cycle 2, n=3,1,9,9,12,9,12,3: number analyzed (Participants) | 3 | 1 | 9 | 9 | 12 | 9 | 12 | 3
  Cmax, Cycle 2, n=3,1,9,9,12,9,12,3 | 0.07490 (43.7) | 0.2496 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.7805 (44.6) | 2.419 (17.8) | 7.129 (37.2) | 29.87 (16.8) | 86.21 (20.4) | 220.0 (19.5)
  Cmax, Cycle 3, n=3,3,6,7,8,8,12,1: number analyzed (Participants) | 3 | 3 | 6 | 7 | 8 | 8 | 12 | 1
  Cmax, Cycle 3, n=3,3,6,7,8,8,12,1 | 0.06961 (23.1) | 0.2269 (16.0) | 0.5577 (31.4) | 1.614 (90.5) | 7.373 (29.2) | 28.02 (18.4) | 92.25 (23.4) | 377.1 (NA) — Geometric coefficient of variation could not be calculated due to single participant
  Cmax, Cycle 4, n=1,3,1,7,4,8,10,0: number analyzed (Participants) | 1 | 3 | 1 | 7 | 4 | 8 | 10 | 0
  Cmax, Cycle 4, n=1,3,1,7,4,8,10,0 | 0.06740 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.2328 (0.2328) | 0.5677 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 1.565 (133.4) | 4.898 (107.0) | 33.06 (14.7) | 96.86 (25.2) |
  Cmax, Cycle 5, n=0,3,0,5,5,7,8,0: number analyzed (Participants) | 0 | 3 | 0 | 5 | 5 | 7 | 8 | 0
  Cmax, Cycle 5, n=0,3,0,5,5,7,8,0 |  | 0.2095 (56.6) |  | 1.664 (161.3) | 7.427 (31.8) | 34.37 (21.3) | 97.28 (28.5) |
  Cmin, Cycle 1, n=0,0,1,6,12,9,12,3: number analyzed (Participants) | 0 | 0 | 1 | 6 | 12 | 9 | 12 | 3
  Cmin, Cycle 1, n=0,0,1,6,12,9,12,3 |  |  | 1.062 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.1120 (77.4) | 0.5031 (90.6) | 5.971 (77.9) | 15.04 (52.1) | 30.32 (40.1)
  Cmin, Cycle 2, n=0,0,0,2,8,9,12,1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 8 | 9 | 12 | 1
  Cmin, Cycle 2, n=0,0,0,2,8,9,12,1 |  |  |  | 0.2482 (5.2) | 0.6783 (161.3) | 6.887 (33.9) | 22.94 (43.8) | 74.09 (NA) — Geometric coefficient of variation could not be calculated due to single participant
  Cmin, Cycle 3, n=0,0,0,3,4,8,10,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 8 | 10 | 0
  Cmin, Cycle 3, n=0,0,0,3,4,8,10,0 |  |  |  | 0.09191 (148.0) | 0.2505 (667.3) | 7.900 (38.3) | 30.77 (40.4) |
  Cmin, Cycle 4, n=0,0,0,3,5,7,8,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 5 | 7 | 8 | 0
  Cmin, Cycle 4, n=0,0,0,3,5,7,8,0 |  |  |  | 0.1536 (95.4) | 0.4313 (383.9) | 9.882 (31.8) | 32.44 (48.4) |
  Cmin, Cycle 5, n=0,0,0,3,4,5,8,0: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 5 | 8 | 0
  Cmin, Cycle 5, n=0,0,0,3,4,5,8,0 |  |  |  | 0.2912 (42.9) | 0.3995 (407.8) | 9.244 (59.5) | 33.69 (51.6) |

45. Secondary Outcome: Part 2B: Cmax and Cmin of GSK3174998
Description: as for outcome 43
Time Frame: as for outcome 43
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 8 | 7 | 4
Micrograms per milliliter
  Cmax, Cycle 1, n=6,6,4: number analyzed (Participants) | 6 | 6 | 4
  Cmax, Cycle 1, n=6,6,4 | 6.921 (19.1) | 5.717 (17.4) | 7.596 (8.7)
  Cmax, Cycle 2, n=8,7,4 | 6.114 (19.3) | 6.139 (21.9) | 7.398 (12.8)
  Cmax, Cycle 3, n=8,4,2: number analyzed (Participants) | 8 | 4 | 2
  Cmax, Cycle 3, n=8,4,2 | 6.574 (17.3) | 7.066 (27.9) | 6.712 (35.5)
  Cmax, Cycle 4, n=4,3,2: number analyzed (Participants) | 4 | 3 | 2
  Cmax, Cycle 4, n=4,3,2 | 7.352 (22.5) | 7.296 (28.1) | 8.162 (6.8)
  Cmax, Cycle 5, n=2,3,2: number analyzed (Participants) | 2 | 3 | 2
  Cmax, Cycle 5, n=2,3,2 | 10.24 (2.6) | 8.684 (29.5) | 9.160 (14.5)
  Cmin, Cycle 1, n=7,5,4: number analyzed (Participants) | 7 | 5 | 4
  Cmin, Cycle 1, n=7,5,4 | 0.3781 (81.6) | 0.7925 (68.4) | 0.3823 (69.5)
  Cmin, Cycle 2, n=7,3,2: number analyzed (Participants) | 7 | 3 | 2
  Cmin, Cycle 2, n=7,3,2 | 0.3082 (187.9) | 1.092 (123.1) | 0.2857 (552.6)
  Cmin, Cycle 3, n=3,3,2: number analyzed (Participants) | 3 | 3 | 2
  Cmin, Cycle 3, n=3,3,2 | 0.7464 (117.5) | 0.9898 (225.3) | 0.3280 (577.1)
  Cmin, Cycle 4, n=2,3,2: number analyzed (Participants) | 2 | 3 | 2
  Cmin, Cycle 4, n=2,3,2 | 0.6753 (207.0) | 0.6852 (947.6) | 0.6114 (93.9)
  Cmin, Cycle 5, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  Cmin, Cycle 5, n=1,2,2 | 1.714 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 0.2250 (4329.5) | 0.8955 (82.7)

46. Secondary Outcome: Part 2A: Plasma Concentrations of Pembrolizumab at Indicated Time Points
Description: Blood samples for PK analysis of pembrolizumab were collected on Day 1: Pre-dose and within 30 minutes, 24 hours after end of pembrolizumab infusion (EOPI); anytime on Days 8,15; Pre-dose on Days 22, 64, 106.
Time Frame: Day 1: Pre-dose and within 30 minutes, 24 hours after end of pembrolizumab infusion; anytime on Days 8,15; Pre-dose on Days 22, 64, 106
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 10 | 11 | 14 | 12 | 12 | 4
Micrograms per milliliter
  Day 1, predose, n=5,4,7,9,10,7,12,3: number analyzed (Participants) | 5 | 4 | 7 | 9 | 10 | 7 | 12 | 3
  Day 1, predose, n=5,4,7,9,10,7,12,3 | 0.000 (0.0000) | 0.000 (0.0000) | 4.414 (11.6791) | 0.000 (0.0000) | 0.404 (1.2776) | 0.000 (0.0000) | 0.008 (0.0284) | 0.000 (0.0000)
  Day1, 30minutes after EOPI, n=5,1,8,6,8,7,10,4: number analyzed (Participants) | 5 | 1 | 8 | 6 | 8 | 7 | 10 | 4
  Day1, 30minutes after EOPI, n=5,1,8,6,8,7,10,4 | 40.860 (28.8970) | 41.000 (NA) — Standard deviation could not be calculated due to single participant | 72.588 (38.0995) | 62.983 (30.3605) | 59.175 (24.1666) | 75.857 (21.3825) | 66.100 (15.2560) | 65.100 (15.6721)
  Day1, 24hour after EOPI, n=5,4,10,8,10,12,12,4: number analyzed (Participants) | 5 | 4 | 10 | 8 | 10 | 12 | 12 | 4
  Day1, 24hour after EOPI, n=5,4,10,8,10,12,12,4 | 44.140 (10.7050) | 56.675 (17.3734) | 65.230 (21.4209) | 50.463 (19.1378) | 53.810 (32.8301) | 54.442 (17.3552) | 51.842 (16.3551) | 48.900 (15.1969)
  Day 8, n=5,4,10,11,14,12,12,4 | 20.340 (6.0719) | 29.600 (8.7882) | 33.850 (13.1268) | 27.618 (10.6709) | 30.757 (13.6721) | 35.600 (16.0615) | 32.792 (9.0537) | 34.025 (11.7196)
  Day 15, n=5,4,10,9,13,12,11,4: number analyzed (Participants) | 5 | 4 | 10 | 9 | 13 | 12 | 11 | 4
  Day 15, n=5,4,10,9,13,12,11,4 | 14.560 (4.1531) | 21.575 (8.7332) | 25.020 (10.7905) | 21.611 (7.3849) | 21.369 (10.9198) | 26.525 (16.4784) | 25.773 (5.3967) | 25.175 (11.0852)
  Day 22, predose, n=5,3,9,10,11,11,12,3: number analyzed (Participants) | 5 | 3 | 9 | 10 | 11 | 11 | 12 | 3
  Day 22, predose, n=5,3,9,10,11,11,12,3 | 12.192 (3.4140) | 12.333 (1.5177) | 17.610 (9.7207) | 17.892 (6.6164) | 18.245 (12.8696) | 19.336 (13.4661) | 18.067 (5.2824) | 18.567 (10.6679)
  Day 64, predose, n=3,3,2,6,5,8,10,0: number analyzed (Participants) | 3 | 3 | 2 | 6 | 5 | 8 | 10 | 0
  Day 64, predose, n=3,3,2,6,5,8,10,0 | 22.433 (6.7678) | 30.133 (8.5008) | 38.550 (13.9300) | 26.560 (14.4486) | 30.720 (8.1940) | 37.000 (14.0108) | 33.640 (11.8732) |
  Day 106, predose, n=1,1,0,6,5,5,8,0: number analyzed (Participants) | 1 | 1 | 0 | 6 | 5 | 5 | 8 | 0
  Day 106, predose, n=1,1,0,6,5,5,8,0 | 18.500 (NA) — Standard deviation could not be calculated due to single participant | 28.100 (NA) — Standard deviation could not be calculated due to single participant |  | 40.150 (14.0395) | 45.420 (20.7985) | 41.400 (17.4579) | 42.850 (17.0662) |

47. Secondary Outcome: Part 2B: Plasma Concentrations of Pembrolizumab at Indicated Time Points
Description: Blood samples for PK analysis of pembrolizumab were collected on Day 1: Pre-dose and within 30 minutes, 24 hours after EOPI; anytime on Days 8,15; Pre-dose on Days 22, 64, 106.
Time Frame: as for outcome 46
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 8 | 5
Micrograms per milliliter
  Day 1, predose, n=8,8,5: number analyzed (Participants) | 8 | 8 | 5
  Day 1, predose, n=8,8,5 | 3.341 (5.7855) | 0.000 (0.0000) | 11.940 (7.3057)
  Day1, 30minutes after EOPI, n=8,6,3: number analyzed (Participants) | 8 | 6 | 3
  Day1, 30minutes after EOPI, n=8,6,3 | 58.650 (12.5860) | 66.600 (15.4104) | 68.633 (7.2473)
  Day1, 24hour after EOPI, n=8,5,0: number analyzed (Participants) | 8 | 5 | 0
  Day1, 24hour after EOPI, n=8,5,0 | 46.800 (12.7711) | 49.960 (7.3228) |
  Day 8, n=9,8,5 | 24.178 (10.0888) | 26.125 (7.6333) | 33.800 (7.5931)
  Day 15, n=9,7,5: number analyzed (Participants) | 9 | 7 | 5
  Day 15, n=9,7,5 | 18.800 (8.8255) | 19.343 (7.3968) | 25.280 (5.7712)
  Day 22, predose, n=9,7,4: number analyzed (Participants) | 9 | 7 | 4
  Day 22, predose, n=9,7,4 | 13.458 (6.4173) | 15.180 (6.4652) | 18.775 (4.7479)
  Day 64, predose, n=4,3,3: number analyzed (Participants) | 4 | 3 | 3
  Day 64, predose, n=4,3,3 | 23.775 (8.2754) | 43.900 (12.1520) | 22.800 (6.0902)
  Day 106, predose, n=2,3,3: number analyzed (Participants) | 2 | 3 | 3
  Day 106, predose, n=2,3,3 | 23.750 (10.6773) | 44.200 (24.5514) | 23.867 (10.1535)

48. Secondary Outcome: Part 2A: AUC(0-tau) of Pembrolizumab
Description: Blood samples for PK analysis of pembrolizumab were collected on Cycle 1 Day 1: Pre-dose and within 30 minutes, 24 hours after EOPI; anytime on Days 8,15, Pre-dose on Day 22 (each dosing cycle was of 21 days). PK parameters of pembrolizumab were calculated using non-compartmental methods.
Time Frame: Cycle 1 Day 1: Pre-dose and within 30 minutes, 24 hours after end of pembrolizumab infusion; anytime on Days 8,15, Pre-dose on Day 22 (each dosing cycle was of 21 days)
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed. There were not enough PK sampling in Cycles 3 and 5 to allow calculation of AUC (0-tau).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 5 | 8 | 8 | 11 | 11 | 3
Day*micrograms per milliliter | 402.11 (43.3) | 561.35 (34.2) | 616.43 (43.7) | 581.61 (34.1) | 528.06 (33.4) | 639.86 (44.8) | 657.22 (22.5) | 703.61 (27.1)

49. Secondary Outcome: Part 2B: AUC(0-tau) of Pembrolizumab
Description: as for outcome 48
Time Frame: as for outcome 48
Population: as for outcome 48
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 6 | 6 | 1
Day*micrograms per milliliter | 470.80 (31.5) | 546.97 (29.1) | 487.40 (NA) — Geometric coefficient of variation could not be calculated due to single participant

50. Secondary Outcome: Part 2A: Cmax of Pembrolizumab
Description: as for outcome 48
Time Frame: as for outcome 48
Population: Pharmacokinetic Population. Only those participants with data available at the indicated data points were analyzed. Post-dose samples were collected in Cycle 1 only and were not collected in Cycles 3 and 5 to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 1 | 6 | 6 | 7 | 7 | 10 | 4
Micrograms per milliliter | 51.83 (48.5) | 41.00 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 79.00 (34.8) | 57.00 (52.7) | 60.20 (36.2) | 72.73 (34.2) | 64.66 (22.0) | 63.65 (25.1)

51. Secondary Outcome: Part 2B: Cmax of Pembrolizumab
Description: as for outcome 48
Time Frame: as for outcome 48
Population: as for outcome 50
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 6 | 6 | 1
Micrograms per milliliter | 56.03 (19.6) | 65.32 (21.1) | 64.60 (NA) — Geometric coefficient of variation could not be calculated due to single participant

52. Secondary Outcome: Part 2A: Cmin of Pembrolizumab
Description: Blood samples for PK analysis of pembrolizumab were collected on Cycle 1 Day 1: Pre-dose and within 30 minutes, 24 hours after EOPI; anytime on Days 8,15; Pre-dose on Days 22; Cycle 3 (Day 64), Cycle 5 (Day 106) (each dosing cycle was of 21 days). PK parameters of pembrolizumab were calculated using non-compartmental methods.
Time Frame: Cycle 1 Day 1: Pre-dose and within 30 minutes, 24 hours after end of pembrolizumab infusion; anytime on Days 8,15; Pre-dose on Days 22; Cycle 3 (Day 64), Cycle 5 (Day 106) (each dosing cycle was of 21 days)
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 3 | 9 | 10 | 11 | 11 | 12 | 3
Micrograms per milliliter
  Cycle 1, n=5,3,9,10,11,11,12,3 | 11.85 (26.8) | 12.27 (12.6) | 15.52 (56.6) | 16.70 (42.6) | 15.81 (54.5) | 16.86 (52.2) | 17.39 (29.6) | 16.78 (57.6)
  Cycle 3, n=3,3,2,6,5,8,10,0: number analyzed (Participants) | 3 | 3 | 2 | 6 | 5 | 8 | 10 | 0
  Cycle 3, n=3,3,2,6,5,8,10,0 | 21.71 (32.7) | 29.40 (27.1) | 37.27 (38.3) | 22.06 (85.1) | 29.93 (25.3) | 34.41 (44.6) | 32.02 (33.2) |
  Cycle 5, n=1,1,0,6,5,5,8,0: number analyzed (Participants) | 1 | 1 | 0 | 6 | 5 | 5 | 8 | 0
  Cycle 5, n=1,1,0,6,5,5,8,0 | 18.50 (NA) — Geometric coefficient of variation could not be calculated due to single participant | 28.10 (NA) — Geometric coefficient of variation could not be calculated due to single participant |  | 37.73 (42.2) | 41.02 (57.0) | 38.13 (49.7) | 39.38 (49.6) |

53. Secondary Outcome: Part 2B: Cmin of Pembrolizumab
Description: as for outcome 52
Time Frame: as for outcome 52
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 7 | 4
Micrograms per milliliter
  Cycle 1, n=9,7,4 | 12.30 (45.9) | 13.88 (50.3) | 18.22 (30.3)
  Cycle 3, n=4,3,3: number analyzed (Participants) | 4 | 3 | 3
  Cycle 3, n=4,3,3 | 22.78 (34.2) | 42.86 (26.9) | 22.28 (26.6)
  Cycle 5, n=2,3,3: number analyzed (Participants) | 2 | 3 | 3
  Cycle 5, n=2,3,3 | 22.52 (49.2) | 39.78 (61.3) | 22.52 (43.1)

54. Secondary Outcome: Part 1: Number of Participants With Positive Antidrug Antibodies (ADAs) Against GSK3174998
Description: Serum samples were collected for the determination of anti-GSK3174998 antibodies using binding ADA assay method using a tiered testing schema: screening, confirmation and titration steps. The presence of treatment emergent ADA was determined using a GSK3174998 bridging style ADA assay with a bio-analytically determined cut-point determined during assay validation. Samples taken after dosing with GSK3174998 that had a value at or above the cut-point was considered treatment-emergent ADA-positive. These ADA positive samples were further evaluated in a confirmatory assay, and confirmed positive samples were further characterized by assessment of titer. Number of participants with confirmed positive anti-GSK3174998 antibodies results at any visit during the study have been presented.
Time Frame: Up to maximum 39 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 8 | 10 | 10 | 4 | 7 | 4
Participants | 0 | 0 | 6 | 7 | 4 | 2 | 2 | 0

55. Secondary Outcome: Part 2A: Number of Participants With Positive ADAs Against GSK3174998
Description: Serum samples were collected for the determination of anti-GSK3174998 antibodies using binding ADA assay method using a tiered testing schema: screening, confirmation and titration steps. The presence of treatment emergent ADA was determined using a GSK3174998 bridging style ADA assay with a bio-analytically determined cut-point (determined during assay validation). Samples taken after dosing with GSK3174998 that had a value at or above the cut-point was considered treatment-emergent ADA-positive. These ADA positive samples were further evaluated in a confirmatory assay, and confirmed positive samples were further characterized by assessment of titer. Number of participants with confirmed positive anti-GSK3174998 antibodies results at any visit during the study have been presented.
Time Frame: Up to maximum 105 weeks
Population: All Treated Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 5 | 9 | 12 | 14 | 12 | 12 | 4
Participants | 2 | 2 | 6 | 8 | 5 | 4 | 0 | 0

56. Secondary Outcome: Part 2B: Number of Participants With Positive ADAs Against GSK3174998
Description: as for outcome 55
Time Frame: Up to maximum 33 weeks
Population: All Treated Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 9 | 7 | 5
Participants | 4 | 1 | 1

57. Secondary Outcome: Part 2A: Number of Participants With Positive ADAs Against Pembrolizumab
Description: Serum samples were collected for the determination of anti-pembrolizumab antibodies using binding ADA assay method using a tiered testing schema: screening, confirmation and titration steps. The presence of treatment emergent ADA was determined using a pembrolizumab bridging style ADA assay with a bio-analytically determined cut-point (determined during assay validation). Samples taken after dosing with pembrolizumab that had a value at or above the cut-point was considered treatment-emergent ADA-positive. These ADA positive samples were further evaluated in a confirmatory assay, and confirmed positive samples were further characterized by assessment of titer. Number of participants with confirmed positive anti-pembrolizumab antibodies results at any visit during the study have been presented.
Time Frame: Up to maximum 105 weeks
Population: All Treated Population. Only those participants with data available at the indicated data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 9 | 10 | 9 | 11 | 8 | 3
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Part 2B: Number of Participants With Positive ADAs Against Pembrolizumab
Description: Serum samples were planned to be collected for the determination of anti-pembrolizumab antibodies using binding ADA assay method using a tiered testing schema: screening, confirmation and titration steps.
Time Frame: Up to maximum 33 weeks
Population: All Treated Population. Data for this outcome measure was not collected as ADA samples were not collected in Part 2B.
Arm/Group | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 39 weeks in Part 1; Up to 105 weeks in Part 2A; Up to 33 weeks in Part 2B
Description: All-cause mortality, SAEs and non-SAEs were collected for All Treated Population which comprised of all participants who received at least one dose of GSK3174998.
Arm/Group | Part 1: GSK3174998 0.003 mg/kg | Part 1: GSK3174998 0.01 mg/kg | Part 1: GSK3174998 0.03 mg/kg | Part 1: GSK3174998 0.1 mg/kg | Part 1: GSK3174998 0.3 mg/kg | Part 1: GSK3174998 1.0 mg/kg | Part 1: GSK3174998 3.0 mg/kg | Part 1: GSK3174998 10.0 mg/kg | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg | Part 2B: Melanoma Cohort | Part 2B: Soft Tissue Sarcoma Cohort | Part 2B: NSCLC Cohort
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 6/8 | 9/10 | 6/10 | 2/4 | 5/7 | 2/4 | 4/5 | 4/5 | 7/10 | 9/12 | 9/14 | 6/12 | 5/12 | 4/4 | 6/9 | 4/8 | 2/5
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 3/8 | 7/10 | 2/10 | 1/4 | 2/7 | 1/4 | 1/5 | 1/5 | 6/10 | 4/12 | 4/14 | 4/12 | 2/12 | 2/4 | 1/9 | 2/8 | 1/5
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 8/8 | 10/10 | 10/10 | 4/4 | 7/7 | 4/4 | 5/5 | 5/5 | 10/10 | 12/12 | 13/14 | 12/12 | 12/12 | 4/4 | 9/9 | 8/8 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3174998 0.003 mg/kg (N=1) | Part 1: GSK3174998 0.01 mg/kg (N=1) | Part 1: GSK3174998 0.03 mg/kg (N=8) | Part 1: GSK3174998 0.1 mg/kg (N=10) | Part 1: GSK3174998 0.3 mg/kg (N=10) | Part 1: GSK3174998 1.0 mg/kg (N=4) | Part 1: GSK3174998 3.0 mg/kg (N=7) | Part 1: GSK3174998 10.0 mg/kg (N=4) | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg (N=5) | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg (N=5) | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg (N=10) | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg (N=14) | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg (N=4) | Part 2B: Melanoma Cohort (N=9) | Part 2B: Soft Tissue Sarcoma Cohort (N=8) | Part 2B: NSCLC Cohort (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pituitary haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to pituitary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3174998 0.003 mg/kg (N=1) | Part 1: GSK3174998 0.01 mg/kg (N=1) | Part 1: GSK3174998 0.03 mg/kg (N=8) | Part 1: GSK3174998 0.1 mg/kg (N=10) | Part 1: GSK3174998 0.3 mg/kg (N=10) | Part 1: GSK3174998 1.0 mg/kg (N=4) | Part 1: GSK3174998 3.0 mg/kg (N=7) | Part 1: GSK3174998 10.0 mg/kg (N=4) | Part 2A: GSK3174998 0.003 mg/kg + Pembrolizumab 200 mg (N=5) | Part 2A: GSK3174998 0.01 mg/kg + Pembrolizumab 200 mg (N=5) | Part 2A: GSK3174998 0.03 mg/kg + Pembrolizumab 200 mg (N=10) | Part 2A: GSK3174998 0.1 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 0.3 mg/kg + Pembrolizumab 200 mg (N=14) | Part 2A: GSK3174998 1.0 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 3.0 mg/kg + Pembrolizumab 200 mg (N=12) | Part 2A: GSK3174998 10.0 mg/kg + Pembrolizumab 200 mg (N=4) | Part 2B: Melanoma Cohort (N=9) | Part 2B: Soft Tissue Sarcoma Cohort (N=8) | Part 2B: NSCLC Cohort (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 3 (4) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (7) | 5 (5) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (11) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 4 (8) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 4 (4) | 5 (6) | 3 (3) | 4 (6) | 1 (1) | 4 (6) | 2 (2) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT02528357/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT02528357/SAP_001.pdf